CLINICAL TRIAL: NCT04334161
Title: Deciphering the Enigma of Postprandial Hyperinsulinaemic Hypoglycaemia After Bariatric Surgery Part 1 B: Evaluation of the Neuro-endocrine Response to Hypoglycaemia.
Brief Title: Evaluation of the Neuro-endocrine Response to Post-prandial Hyperinsulinaemic Hypoglycaemia.
Acronym: DEEP1B
Status: Completed | Type: Observational
Sponsor: Lia Bally (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Professor, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: DEEP1B
Record Dates: First submitted 2020-03-30; First posted 2020-04-06 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Roux-en-y Gastric Bypass; Post Prandial Hypoglycemia
Keywords: Counter-regulation to hypoglycemia; Neuro-endocrine response; Glucagon
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PHH patients: Patients with Roux-en-Y gastric bypass ≥1 year ago and confirmed postprandial hyperglycaemic hypoglycaemia (PHH). PHH is defined as postprandial plasma or sensor glucose<3.0mmol/l according to the International Hypoglycaemia Study Group and exclusion of other causes of hypoglycaemia
  Interventions: Combination Product: Administration of glucose and controlled induction of hypoglycaemia.
- non-PHH gastric bypass patients: Patients with Roux-en-Y gastric bypass ≥1 year ago without evidence of PHH.
  Interventions: Combination Product: Administration of glucose and controlled induction of hypoglycaemia.
- non-PHH sleeve gastrectomy patients: Patients with sleeve gastrectomy ≥1 year ago without evidence PHH.
  Interventions: Combination Product: Administration of glucose and controlled induction of hypoglycaemia.
- non-PHH non-surgical controls: Absence of any conditions or previous surgery known to affect gastro-intestinal integrity and food absorption.
  Interventions: Combination Product: Administration of glucose and controlled induction of hypoglycaemia.

INTERVENTIONS:
Combination Product: Administration of glucose and controlled induction of hypoglycaemia. — Functional metabolic test involving a 15g oral glucose load (enriched with 1.5% U-13C glucose) and subsequent controlled 20min hypoglycaemic clamp period. Neuroendocrine response will be assessed using frequent blood samples for hormones and metabolites, continuous heart rate monitoring and evaluation for hypoglycaemic symptoms.

SUMMARY:
The primary objective of this study is to assess the neuro-endocrine response to hypoglycaemia in PHH vs. non-PHH post-gastric bypass individuals.

DETAILED DESCRIPTION:
Obesity is a major global public health concern, for which the most effective therapy is bariatric surgery. Beyond weight loss, bariatric surgery exerts powerful effects on glucose metabolism, achieving complete type 2 diabetes remission in up to 70% of cases. An exaggeration of these effects, however, can result in an increasingly recognized metabolic complication known as postprandial hyperinsulinaemic hypoglycaemia (PHH). The condition manifests 1-3 years after surgery with hypoglycaemic episodes after meals. Emerging data suggest that PHH is more frequent than previously thought and affects approximately 30% of postoperative patients, more commonly after gastric bypass than sleeve gastrectomy . Despite such frequency, the underlying pathophysiology of PHH remains incompletely understood.

A striking finding in PHH patients is the observed lack of insulin suppression and inadequate glucagon response to the sharply falling glucose levels. The blunted glucagon response to hypoglycaemia may result from altered alpha-cell function (acute or chronic) and an interaction with gut hormones (e.g. glucagon-like peptide 1 (GLP-1) that is known to exert glucagon-inhibitory effects) or altered brain signalling. It is conceivable that, both, lack of endogenous insulin suppression in response to falling postprandial blood glucose levels and impaired glucagon secretion contribute to PHH.

Further neuroendocrine regulatory processes to counteract hypoglycaemia involve catecholamines, cortisol, growth hormone and autonomic nervous system activity. Two previous studies examined counter-regulatory hormones during experimentally induced hypoglycaemia in patients after gastric bypass surgery and found lower levels than before surgery, suggesting that bariatric surgery per se influences counter-regulation to hypoglycaemia. Underlying mechanisms remain speculative. Of note, impaired neuroendocrine counter-regulation to hypoglycaemia is further supported by the high proportion of asymptomatic patients, which may be reflective of impaired hypoglycaemia awareness. The role of counter-regulatory hormones in PHH patients remains not fully understood.

Apart from the neuroendocrine milieu, effectiveness of hypoglycaemia counter-regulation depends on the capacity to provide glucose from the liver, also known as endogenous glucose production. In healthy humans, approximately 85% of the glucose produced by the liver during the initial 60-90min of hypoglycaemia is derived from liver glycogen. Postprandial hepatic glycogen stores, in turn, depend heavily on the hepatic glucose uptake following a meal. Postprandial hepatic glucose disposal and mobilization of hepatic glucose during hypoglycaemia in PHH patients remain unexplored to date.

There is currently no evidence, that increased insulin sensitivity is implicated in the pathophysiology of PHH. Conversely, previous studies suggested increased non-insulin dependent whole body glucose uptake in PHH compared to non-PHH in the light of similar or even decreased insulin sensitivity.

The primary objective of this study is to assess the neuro-endocrine response to hypoglycaemia in PHH vs. non-PHH post-gastric bypass individuals. The investigators hypothesize that the glucagon response to standardized and controlled hypoglycaemia is significantly diminished in PHH vs. non-PHH post-gastric bypass individuals. Involvement of non-surgical non-PHH controls and sleeve-gastrectomy non-PHH controls will allow to explore effects of bariatric surgery on counter-regulatory mechanisms to hypoglycaemia, including differences between procedures (gastric bypass vs. sleeve gastrectomy).

ELIGIBILITY:
Inclusion criteria for PHH patients (Group 1):

* Aged ≥18 years
* Roux-en-Y gastric bypass ≥1 year ago
* PHH defined as postprandial plasma or sensor glucose<3.0mmol/l according to the International Hypoglycaemia Study Group (1) and exclusion of other causes of hypoglycaemia

Inclusion criteria for non-PHH surgical controls (Group 2 and 3):

* Aged ≥18 years
* Roux-en-Y gastric bypass (Group 2) or sleeve gastrectomy (Group 3) ≥1 year ago
* No evidence of PHH

Inclusion criteria for non-PHH non-surgical controls (Group 4):

* Aged ≥18 years
* Absence of any condition or previous surgery known to affect gastro-intestinal integrity and food absorption

Exclusion criteria for all Groups:

* Clinically relevant weight changes (≥5%) within the past 3 months
* Incapacity to give informant consent
* Historical or current diabetes based on HbA1c ≥6.5% without glucose-lowering treatment
* Haemoglobin level below 13.5 g/l
* Ongoing treatment with glucose-lowering drugs, anorectic drugs, steroids or any medications known to affect gastric motility
* Active heart, lung, liver, gastrointestinal, renal or neurological disease
* Inability to follow study procedures
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited by referral from our outpatient endocrine clinic and collaborating Centres of Excellence for Metabolic Surgery. Non-surgical controls will be recruited through advertisement according to guidelines from swissethics.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Glucagon response during the 20min hypoglycaemic period as defined using the area under the concentration curve (AUC) | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)

SECONDARY OUTCOMES:
Response of C-peptide during the 20min hypoglycaemic period as determined by the area under the curve (AUC). | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)
Response of cortisol during the 20min hypoglycaemic period as determined by the area under the curve (AUC). | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)
Response of adrenaline during the 20min hypoglycaemic period as determined by the area under the curve (AUC). | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)
Response of noradrenaline during the 20min hypoglycaemic period as determined by the area under the curve (AUC). | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)
Response of growth hormone during the 20min hypoglycaemic period as determined by the area under the curve (AUC). | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)
Response of Glucagon-like peptide (GLP-1) during the 20min hypoglycaemic period as determined by the area under the curve (AUC). | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)
Response of glucose-dependent insulinotropic polypeptide (GIP) during the 20min hypoglycaemic period as determined by the area under the curve (AUC). | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)
Response of peptide tyrosine tyrosine (PYY) during the 20min hypoglycaemic period as determined by the area under the curve (AUC). | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)
Response of pancreatic polypeptide (PP) during the 20min hypoglycaemic period as determined by the area under the curve (AUC). | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)
Endogenous glucose production during the 20min hypoglycaemic period as defined using the AUC of the rate of endogenous glucose production (Total rate of glucose appearance-Rate of glucose infusion) | 20 minutes of the hypoglycaemic period (from 150 to 170 minutes after the oral glucose load)

OTHER OUTCOMES:
Time course of the hormonal response during the whole experiment. | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
  Assessed hormones: insulin, C-peptide, glucagon, cortisol, adrenaline, noradrenaline, Growth Hormone, Glucagon-like peptide 1 [GLP-1], glucose-dependent insulinotropic polypeptide [GIP], peptide tyrosine tyrosine [PYY], pancreatic polypeptide [PP]
Time course of rate of glucose appearance (Ra total) during the whole experiment | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Time course of rate of glucose disappearance (Rd) during the whole experiment | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Time course of rate of meal-derived glucose appearance (Ra oral) during the whole experiment | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Time course of rate of endogenous glucose production (EGP) during the whole experiment | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Total beta-cell function (total beta-cell glucose responsiveness) | Calculated from time of the oral glucose load (T0) to 120 minutes after the oral glucose load (T120)
  Calculated from the oral c-peptide minimal model
Dynamic beta-cell function (dynamic beta-cell glucose responsiveness) | Calculated from time of the oral glucose load (T0) to 120 minutes after the oral glucose load (T120)
  Calculated from the oral c-peptide minimal model
Static beta-cell function indices (static beta-cell glucose responsiveness) | Calculated from time of the oral glucose load (T0) to 120 minutes after the oral glucose load (T120)
  Calculated from the oral c-peptide minimal model
Insulin clearance | Calculated from time of the oral glucose load (T0) to 120 minutes after the oral glucose load (T120)
  Calculated using the oral minimal model
Hepatic insulin extraction | Calculated from time of the oral glucose load (T0) to 120 minutes after the oral glucose load (T120)
  Calculated using the oral minimal model
Heart rate in response to the meal and during hypoglycaemia | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Heart rate variability (low to high frequency power ratio) in response to the meal and during hypoglycaemia | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Heart rate variability (high frequency power) in response to the meal and during hypoglycaemia | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Heart rate variability (low frequency power) in response to the meal and during hypoglycaemia | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Systolic blood pressure in response to the meal and during hypoglycaemia | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Diastolic blood pressure in response to the meal and during hypoglycaemia | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Time course of haematocrit during the whole experiment | From the start of the experiment (100 minutes before the oral glucose load) until the end of the experiment (170 minutes after the oral glucose load)
Autonomous symptoms in response to the meal and during hypoglycaemia according to the Edinburgh Hypoglycaemia Scale. | 40 minutes after the oral glucose load
  Sum of the scores of the autonomous symptoms from the Edinburgh hypoglycemia Scale. Each score is based on the patient's evaluation of the respective symptom using a Likert scale (1-7). A higher score means a more intense hypoglycaemia feeling.
Autonomous symptoms in response to the meal and during hypoglycaemia according to the Edinburgh Hypoglycaemia Scale. | 100 minutes after the oral glucose load
  Sum of the scores of the autonomous symptoms from the Edinburgh hypoglycemia Scale. Each score is based on the patient's evaluation of the respective symptom using a Likert scale (1-7). A higher score means a more intense hypoglycaemia feeling.
Autonomous symptoms in response to the meal and during hypoglycaemia according to the Edinburgh Hypoglycaemia Scale. | 140 minutes after the oral glucose load
  Sum of the scores of the autonomous symptoms from the Edinburgh hypoglycemia Scale. Each score is based on the patient's evaluation of the respective symptom using a Likert scale (1-7). A higher score means a more intense hypoglycaemia feeling.
Neuroglycopenic symptoms in response to the meal and during hypoglycaemia according to the Edinburgh Hypoglycaemia Scale. | 40 minutes after the oral glucose load
  Sum of the scores of the neuroglycopenic symptoms from the Edinburgh hypoglycemia Scale. Each score is based on the patient's evaluation of the respective symptom using a Likert scale (1-7). A higher score means a more intense hypoglycaemia feeling.
Neuroglycopenic symptoms in response to the meal and during hypoglycaemia according to the Edinburgh Hypoglycaemia Scale. | 100 minutes after the oral glucose load
  Sum of the scores of the neuroglycopenic symptoms from the Edinburgh hypoglycemia Scale. Each score is based on the patient's evaluation of the respective symptom using a Likert scale (1-7). A higher score means a more intense hypoglycaemia feeling.
Neuroglycopenic symptoms in response to the meal and during hypoglycaemia according to the Edinburgh Hypoglycaemia Scale. | 140 minutes after the oral glucose load
  Sum of the scores of the neuroglycopenic symptoms from the Edinburgh hypoglycemia Scale. Each score is based on the patient's evaluation of the respective symptom using a Likert scale (1-7). A higher score means a more intense hypoglycaemia feeling.

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD, PhD, Principal Investigator — University Hospital Bern & University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tripyla A, Herzig D, Reverter-Branchat G, Pavan J, Schiavon M, Eugster PJ, Grouzmann E, Nakas CT, Sauvinet V, Meiller L, Zehetner J, Giachino D, Nett P, Gawinecka J, Del Favero S, Thomas A, Thevis M, Dalla Man C, Bally L. Counter-regulatory responses to postprandial hypoglycaemia in patients with post-bariatric hypoglycaemia vs surgical and non-surgical control individuals. Diabetologia. 2023 Apr;66(4):741-753. doi: 10.1007/s00125-022-05861-9. Epub 2023 Jan 17. PMID 36648553